CLINICAL TRIAL: NCT06329219
Title: Water-filtered Infrared-A Radiation in Patients With Hand Osteoarthritis - a Randomized Controlled Trial
Brief Title: Water-filtered Infrared-A Radiation in Patients With Hand Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: wIRA
Record Dates: First submitted 2024-03-19; First posted 2024-03-25 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Hand Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiation (Experimental): Participants in the intervention group each receive a hyperthermia device for water-filtered Infrared-A radiation.
  Interventions: Device: water-filtered Infrared-A radiation
- Waiting list (No Intervention): Participants in the control group initially receive no therapeutic intervention, but can receive it after the study's last visit for 3 months.

INTERVENTIONS:
Device: water-filtered Infrared-A radiation — The water-filtered Infrared-A radiation device is designed for self-administered home treatments. The regimen prescribes 30-minute sessions, five times weekly, spanning 12 weeks.
  Arms: Radiation

SUMMARY:
The aim of this clinical trial is to evaluate the effects of water-filtered Infrared-A radiation on patients suffering from hand osteoarthritis. The main questions it aims to answer are:

* Does water-filtered Infrared-A radiation reduce pain and improve the function of finger joints over time?
* Are patients satisfied with the treatment results when compared to those who were on a wait-list?

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of finger polyarthritis (confirmed by a specialist, radiological findings available)
* Local pain for more than 50% of the day in the past 3 months.
* Subjective pain intensity of local pain in the last 24 hours on a VAS scale of 0 to 10 being >4.
* No planned local treatment in the next 6 months.
* No planned intra-articular injections within the next 6 months.
* The patient must be able to understand the study explanations and appropriately follow the instructions of the investigating physician.

Exclusion Criteria:

* Chronic inflammatory joint diseases.
* Poor general health.
* Febrile diseases.
* Fibromyalgia syndrome.
* Psychotic disorders.
* Severe comorbidities.
* Acute unclear skin diseases.
* Heat urticaria.
* Painful diseases/diagnoses of the shoulder and/or arm.
* Lymphatic vessel diseases (lymphedema, lymphangitis).
* Porphyria.
* Pain-associated diseases/diagnoses of the shoulder and/or arm.
* Intra-articular injections or arthroscopies within the last 3 months.
* Previous or planned surgical procedure on the affected joints in the last 8 weeks or in the upcoming 6 months.
* Intake or application of photosensitizing drugs or extracts (e.g., porphyrins, tetracyclines, sulfonamides, psoralenes, St. John's wort).
* Systemic medication with glucocorticoids or immunosuppressants.
* Pain medication with opioid analgesics.
* Known pregnancy.
* Concurrent participation in another clinical trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pain in the finger joints on visual analogue scale | Baseline, 12 weeks
  Average pain in the finger joints over the last 7 days after 12 weeks compared to baseline on the Visual Analog Scale (VAS, 0-100mm) compared to the waiting list control group.

SECONDARY OUTCOMES:
Hand Dynamometer | Baseline, 6 weeks, 12 weeks, 24 weeks
  Grip strength measured using a Hand Dynamometer (SAEHAN Corporation)
Disabilities of Arm, Shoulder and Hand (DASH) questionnaire | Baseline, 6 weeks, 12 weeks, 24 weeks
  Assessing full scale, range 0-100, higher score meaning a better outcome
Pain Self-Efficacy Questionnaire | Baseline, 6 weeks, 12 weeks, 24 weeks
  Assessing full scale, range 0-100, higher score meaning a better outcome
Hospital Anxiety and Depression Scale (HADS) | Baseline, 6 weeks, 12 weeks, 24 weeks
  Assessing full scale, range 0-100, higher score meaning a better outcome
Short Form (SF)-36 Health Survey (SF-36) | Baseline, 6 weeks, 12 weeks, 24 weeks
  Assessing full scale, range 0-100, higher score meaning a better outcome
Functional Index for Hand OsteoArthritis (FIHOA) | Baseline, 6 weeks, 12 weeks, 24 weeks
  Assessing functional impairment, scoring from 0 (no functional impairment) to 30 points (maximal impairment).
Tolerability of the intervention | Baseline, 6 weeks, 12 weeks, 24 weeks
  Monitoring tolerability of the intervention (5-point Likert scale, 1=very good tolerability to 5=very bad tolerability)
Pain medication (number per day) | Baseline, 6 weeks, 12 weeks, 24 weeks
  Documenting changes in pain medication and pain medication on demand

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, Principal Investigator — Charite University, Berlin, Germany; Rainer Stange, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin at the Department of Internal and Integrative Medicine, Immanuel Krankenhaus Berlin, Wannsee, State of Berlin, Germany